CLINICAL TRIAL: NCT02429388
Title: High-Dose Aldactone for Treatment of Diuretic Resistant Heart Failure
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Principal Investigator left institution prior to subjects being enrolled
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20140274H
Record Dates: First submitted 2014-09-27; First posted 2015-04-29 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Heart Failure
Keywords: Heart failure; Spironolactone; Diuretics
MeSH Terms: conditions — Heart Failure | interventions — Spironolactone; Sodium Channel Blockers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High dose spironolactone (Experimental): This arm of the study will include addition of high dose spironolactone upto 100mg twice daily in adjunct to usual care of hospitalized acute decompensated heart failure patients with loop diuretics.
  Interventions: Drug: Spironolactone
- Usual Care (No Intervention): This arm of the study will continue the usual care of hospitalized acute decompensated heart failure patients with loop diuretics.

INTERVENTIONS:
Drug: Spironolactone — Administration of spironolactone 25-50mg orally twice daily for two days and subsequently titrated upto 100mg twice daily with daily serum potassium monitoring. Spironolactone will continue until patient is euvolemic and appropriate for discharge. Titration of loop diuretics in this arm will not be escalated.
  Other Names: aldactone; potassium-sparing diuretics
  Arms: High dose spironolactone

SUMMARY:
Prospective, open-label, randomized cohort study comparing adding high-dose spironolactone to usual heart failure care versus usual care in patients with acute decompensated heart failure. Patients will be randomized in a 1:1 fashion to either usual care or high-dose spironolactone plus usual care. Both arms of the study will continue with treatment of ADHF until euvolemia as defined as the resolution of pulmonary edema, peripheral edema, abdominal bloating and/or jugular venous distention. Assessment of clinical status and serum electrolytes, symptoms and renal function will be performed in accordance to standard of care.

DETAILED DESCRIPTION:
Congestive heart failure (CHF) is common and currently affects an estimated 6.6 million adults in the United States (1). In addition being highly prevalent, CHF is responsible for ~ 1 million hospital discharges per year and approximately 50% of patients with CHF will die within 5 years making it a highly morbid and lethal disease (1).

Manifestations of CHF include symptoms of volume overload such as dyspnea, abdominal bloating and/or fatigue. The genesis of these symptoms begins with loss of the integrity of arterial circulation due to decreased cardiac output (2). Decreased activation of mechanoreceptors in the carotid sinus, left ventricle, aortic arch and renal afferent arterioles due to lower systemic arterial pressure stimulates the sympathetic nervous system (SNS), renal-angiotensin-aldosterone system (RAAS) and non-osmotic release of arginine vasopressin (3). As a result, sodium reabsorption in the proximal tubule followed by water absorption increases causing accumulation of intravascular volume to compensating for arterial underfilling (4). Consequently, activation of neurohumoral reflexes result in increased cardiac afterload and preload, cardiac remodeling, hyponatremia and pulmonary edema (5). Renal vasoconstriction, sodium and water retention leads to a continuous positive feedback loop of further salt and water accumulation accompanied by further renal vasoconstriction (6).

Diuretic therapy is the most common means to relieve congestion in acute decompensated heart failure (ADHF) and approximately 90% of patients are treated with loop diuretics (7). Although loop diuretics are a cornerstone ADHF care and carries the highest level of recommendation by the American Heart Association (Class I); the guideline is supported by the lowest level of evidence (Class C) (8). While effective at natriuresis, loop diuretics are known to stimulate the SNS and RAAS, both of which have adverse consequence in heart failure (9,10). Not only is the RAAS system stimulated due to changes in arterial filling, furosemide blocks sodium chloride transport at the macula densa causing renin release independent of renal sodium loss (11). With increase stimulation of renin release, vasoconstriction of the renal artery ensues causing or further exacerbating renal insufficiency (12). Long-term utilization of loop diuretics results in hypertrophy of the distal nephron and increased expression of a sodium chloride co-transporter (13). These changes along with increased aldosterone levels further enhances distal sodium reabsorption and prevents aldosterone escape (14).

In treating heart failure patients as a population, diuretic resistance is encountered commonly and escalating doses of furosemide may be utilized to achieve fluid loss (15). Clinically, use of high-doses of loop diuretics is associated with greater rates of clinical events such as mechanical ventilation and myocardial infarction compared to low-dose loop diuretics (16). High-dose loop diuretic administration is associated with worsening renal function (17), increased length of hospital stay and greater in-hospital mortality (17-19). There is in fact a linear correlation with diuretic dose and mortality (20).

Given the potential hazards of administering loop diuretics in CHF patients, the remaining options are limited. Changing diuretics strategies from bolus to continuous loop diuretic infusion does not appear to change overall outcomes (21). Alternative strategies for relieving congestion include inhibition of the distal nephron using thiazide diuretics. Thiazide diuretics work synergistically with loop diuretics to induce natriuresis but have an independent association with worsening renal function and death (20,22). Utilizing inotropes to increasing renal perfusion pressure may improve natriuresis, however, it comes with the price of increasing mortality regardless of whether beta-adrenergic agonists (dobutamine) or phosphodiesterase inhibitors are used (23,24). Ultrafiltration and mechanical unloading of the heart is another therapeutic option, however it was found to be ineffective and associated with worsening renal function (25). Even low doses of dopamine or nesiritide were not effective in improving outcomes in patients with cardiorenal syndrome (26). Higher doses of spironolactone were recently shown to be safe in a prospective cohort treated for acute decompensated heart failure (27). Recently a case report was published showing that patients hospitalized with congestive heart failure, worsening renal function and diuretic resistance were able to be diuresed without adverse effect on renal function or hyperkalemia by treating with escalating doses of spironolactone (28)

The study will be a prospective, open-label, randomized cohort study comparing adding high-dose spironolactone to usual heart failure care versus usual care in patients with acute decompensated heart failure. Patients will be randomized in a 1:1 fashion to either usual care or high-dose spironolactone plus usual care. Both arms of the study will continue with treatment of ADHF until euvolemia as defined as the resolution of pulmonary edema, peripheral edema, abdominal bloating and/or jugular venous distention. Assessment of clinical status, urine and serum electrolytes, symptoms and renal function will be performed in accordance to standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older patients with congestive heart failure
2. Hypervolemic by at least 2 of the following criteria: 1) Peripheral edema; 2) jugular venous distention greater than 7 cm; 3) radiographic pulmonary edema or pleural effusion; 4) enlarged liver or ascites; 5) pulmonary rales, paroxysmal nocturnal dyspnea or orthopnea
3. Diuretic resistance as defined by loop diuretic requirements of furosemide greater or equal to 160 mg IV total daily dose or equivalent dose of torsemide or bumetanide. ( 1 mg bumetanide = 10 mg torsemide = 20 mg furosemide)
4. Estimated glomerular filtration rate (eGFR) of > 30ml/min. according to the MDRD Study equation at the time of admission.
5. Female patients of child bearing potential must have a negative urine pregnancy test to be eligible.

Exclusion Criteria:

1. Acute coronary syndrome
2. Patients with a baseline eGFR < 30 ml/min according to the MDRD equation.
3. Baseline potassium serum concentration 5.3 meq/L
4. Requirement for intravenous pressors
5. Systemic infection
6. Patients with concomitant end-stage liver disease
7. Significant valvular disease
8. Patients with pulmonary embolism
9. Patients with high output heart failure
10. Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of adjunctive high-dose Spironolactone on weight loss. | 7 days
  Weight will be tracked from enrollment to 7 days or when patient reaches euvolemia for all patients, whichever occurs first.

SECONDARY OUTCOMES:
Efficacy of adjunctive high-dose Spironolactone on dyspnea. | 7 days
  Using Likert scale, dyspnea and functional status will be assessed at enrollment and re-evaluate at 7days or at euvolemia for all patients, whichever occurs first.
Risk of hyperkalemia and renal dysfunction with use of adjunctive high-dose Spironolactone. | 7 days
  Assessment of serum potassium and creatinine daily on all patients to assess relative safety of spironolactone use in diuretic resistant heart failure patients.
Length of hospitalization | 7 days
  Comparison of length of hospitalization with use of high dose spironolactone to heart failure therapy compared to usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Marvin H Eng, M.D., Principal Investigator — University of Texas Heatlh Science Center at San Antonio
Locations (1):
- University Hospital, San Antonio, Texas, United States

REFERENCES:
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):e2-e220. doi: 10.1161/CIR.0b013e31823ac046. Epub 2011 Dec 15. No abstract available. PMID 22179539
- [Background] Schrier RW, Abraham WT. Hormones and hemodynamics in heart failure. N Engl J Med. 1999 Aug 19;341(8):577-85. doi: 10.1056/NEJM199908193410806. No abstract available. PMID 10451464
- [Background] Schrier RW. Water and sodium retention in edematous disorders: role of vasopressin and aldosterone. Am J Med. 2006 Jul;119(7 Suppl 1):S47-53. doi: 10.1016/j.amjmed.2006.05.007. PMID 16843085
- [Background] Schrier RW. Decreased effective blood volume in edematous disorders: what does this mean? J Am Soc Nephrol. 2007 Jul;18(7):2028-31. doi: 10.1681/ASN.2006111302. Epub 2007 Jun 13. PMID 17568020
- [Background] Hirsch AT, Pinto YM, Schunkert H, Dzau VJ. Potential role of the tissue renin-angiotensin system in the pathophysiology of congestive heart failure. Am J Cardiol. 1990 Oct 2;66(11):22D-30D; discussion 30D-32D. doi: 10.1016/0002-9149(90)90473-e. PMID 2220602
- [Background] Schrier RW, De Wardener HE. Tubular reabsorption of sodium ion: influence of factors other than aldosterone and glomerular filtration rate. 2. N Engl J Med. 1971 Dec 2;285(23):1292-303. doi: 10.1056/NEJM197112022852305. No abstract available. PMID 4398836
- [Background] Adams KF Jr, Fonarow GC, Emerman CL, LeJemtel TH, Costanzo MR, Abraham WT, Berkowitz RL, Galvao M, Horton DP; ADHERE Scientific Advisory Committee and Investigators. Characteristics and outcomes of patients hospitalized for heart failure in the United States: rationale, design, and preliminary observations from the first 100,000 cases in the Acute Decompensated Heart Failure National Registry (ADHERE). Am Heart J. 2005 Feb;149(2):209-16. doi: 10.1016/j.ahj.2004.08.005. PMID 15846257
- [Background] Hunt SA, Abraham WT, Chin MH, Feldman AM, Francis GS, Ganiats TG, Jessup M, Konstam MA, Mancini DM, Michl K, Oates JA, Rahko PS, Silver MA, Stevenson LW, Yancy CW, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Halperin JL, Hiratzka LF, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology; American Heart Association Task Force on Practice Guidelines; American College of Chest Physicians; International Society for Heart and Lung Transplantation; Heart Rhythm Society. ACC/AHA 2005 Guideline Update for the Diagnosis and Management of Chronic Heart Failure in the Adult: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Update the 2001 Guidelines for the Evaluation and Management of Heart Failure): developed in collaboration with the American College of Chest Physicians and the International Society for Heart and Lung Transplantation: endorsed by the Heart Rhythm Society. Circulation. 2005 Sep 20;112(12):e154-235. doi: 10.1161/CIRCULATIONAHA.105.167586. Epub 2005 Sep 13. No abstract available. PMID 16160202
- [Background] Francis GS, Goldsmith SR, Levine TB, Olivari MT, Cohn JN. The neurohumoral axis in congestive heart failure. Ann Intern Med. 1984 Sep;101(3):370-7. doi: 10.7326/0003-4819-101-3-370. PMID 6147109
- [Background] Bayliss J, Norell M, Canepa-Anson R, Sutton G, Poole-Wilson P. Untreated heart failure: clinical and neuroendocrine effects of introducing diuretics. Br Heart J. 1987 Jan;57(1):17-22. doi: 10.1136/hrt.57.1.17. PMID 3541995
- [Background] He XR, Greenberg SG, Briggs JP, Schnermann J. Effects of furosemide and verapamil on the NaCl dependency of macula densa-mediated renin secretion. Hypertension. 1995 Jul;26(1):137-42. doi: 10.1161/01.hyp.26.1.137. PMID 7607716
- [Background] Ellison DH. Diuretic therapy and resistance in congestive heart failure. Cardiology. 2001;96(3-4):132-43. doi: 10.1159/000047397. PMID 11805380
- [Background] Abdallah JG, Schrier RW, Edelstein C, Jennings SD, Wyse B, Ellison DH. Loop diuretic infusion increases thiazide-sensitive Na(+)/Cl(-)-cotransporter abundance: role of aldosterone. J Am Soc Nephrol. 2001 Jul;12(7):1335-1341. doi: 10.1681/ASN.V1271335. PMID 11423562
- [Background] Ellison DH, Velazquez H, Wright FS. Adaptation of the distal convoluted tubule of the rat. Structural and functional effects of dietary salt intake and chronic diuretic infusion. J Clin Invest. 1989 Jan;83(1):113-26. doi: 10.1172/JCI113847. PMID 2910903
- [Background] Bansal S, Lindenfeld J, Schrier RW. Sodium retention in heart failure and cirrhosis: potential role of natriuretic doses of mineralocorticoid antagonist? Circ Heart Fail. 2009 Jul;2(4):370-6. doi: 10.1161/CIRCHEARTFAILURE.108.821199. PMID 19808361
- [Background] Heywood JT, Fonarow GC, Costanzo MR, Mathur VS, Wigneswaran JR, Wynne J; ADHERE Scientific Advisory Committee and Investigators. High prevalence of renal dysfunction and its impact on outcome in 118,465 patients hospitalized with acute decompensated heart failure: a report from the ADHERE database. J Card Fail. 2007 Aug;13(6):422-30. doi: 10.1016/j.cardfail.2007.03.011. PMID 17675055
- [Background] Butler J, Forman DE, Abraham WT, Gottlieb SS, Loh E, Massie BM, O'Connor CM, Rich MW, Stevenson LW, Wang Y, Young JB, Krumholz HM. Relationship between heart failure treatment and development of worsening renal function among hospitalized patients. Am Heart J. 2004 Feb;147(2):331-8. doi: 10.1016/j.ahj.2003.08.012. PMID 14760333
- [Background] Peacock WF, Costanzo MR, De Marco T, Lopatin M, Wynne J, Mills RM, Emerman CL; ADHERE Scientific Advisory Committee and Investigators. Impact of intravenous loop diuretics on outcomes of patients hospitalized with acute decompensated heart failure: insights from the ADHERE registry. Cardiology. 2009;113(1):12-9. doi: 10.1159/000164149. Epub 2008 Oct 17. PMID 18931492
- [Background] Butler J, Chirovsky D, Phatak H, McNeill A, Cody R. Renal function, health outcomes, and resource utilization in acute heart failure: a systematic review. Circ Heart Fail. 2010 Nov;3(6):726-45. doi: 10.1161/CIRCHEARTFAILURE.109.920298. No abstract available. PMID 21081740
- [Background] Forman DE, Butler J, Wang Y, Abraham WT, O'Connor CM, Gottlieb SS, Loh E, Massie BM, Rich MW, Stevenson LW, Young JB, Krumholz HM. Incidence, predictors at admission, and impact of worsening renal function among patients hospitalized with heart failure. J Am Coll Cardiol. 2004 Jan 7;43(1):61-7. doi: 10.1016/j.jacc.2003.07.031. PMID 14715185
- [Background] Felker GM, Lee KL, Bull DA, Redfield MM, Stevenson LW, Goldsmith SR, LeWinter MM, Deswal A, Rouleau JL, Ofili EO, Anstrom KJ, Hernandez AF, McNulty SE, Velazquez EJ, Kfoury AG, Chen HH, Givertz MM, Semigran MJ, Bart BA, Mascette AM, Braunwald E, O'Connor CM; NHLBI Heart Failure Clinical Research Network. Diuretic strategies in patients with acute decompensated heart failure. N Engl J Med. 2011 Mar 3;364(9):797-805. doi: 10.1056/NEJMoa1005419. PMID 21366472
- [Background] Peacock WF 4th, De Marco T, Fonarow GC, Diercks D, Wynne J, Apple FS, Wu AH; ADHERE Investigators. Cardiac troponin and outcome in acute heart failure. N Engl J Med. 2008 May 15;358(20):2117-26. doi: 10.1056/NEJMoa0706824. PMID 18480204
- [Background] Klein L, Massie BM, Leimberger JD, O'Connor CM, Pina IL, Adams KF Jr, Califf RM, Gheorghiade M; OPTIME-CHF Investigators. Admission or changes in renal function during hospitalization for worsening heart failure predict postdischarge survival: results from the Outcomes of a Prospective Trial of Intravenous Milrinone for Exacerbations of Chronic Heart Failure (OPTIME-CHF). Circ Heart Fail. 2008 May;1(1):25-33. doi: 10.1161/CIRCHEARTFAILURE.107.746933. PMID 19808267
- [Background] Applefeld MM, Newman KA, Sutton FJ, Reed WP, Roffman DS, Talesnick BS, Grove WR. Outpatient dobutamine and dopamine infusions in the management of chronic heart failure: clinical experience in 21 patients. Am Heart J. 1987 Sep;114(3):589-95. doi: 10.1016/0002-8703(87)90757-5. PMID 3630900
- [Background] Felker GM, Mentz RJ. Diuretics and ultrafiltration in acute decompensated heart failure. J Am Coll Cardiol. 2012 Jun 12;59(24):2145-53. doi: 10.1016/j.jacc.2011.10.910. PMID 22676934
- [Background] Chen HH, Anstrom KJ, Givertz MM, Stevenson LW, Semigran MJ, Goldsmith SR, Bart BA, Bull DA, Stehlik J, LeWinter MM, Konstam MA, Huggins GS, Rouleau JL, O'Meara E, Tang WH, Starling RC, Butler J, Deswal A, Felker GM, O'Connor CM, Bonita RE, Margulies KB, Cappola TP, Ofili EO, Mann DL, Davila-Roman VG, McNulty SE, Borlaug BA, Velazquez EJ, Lee KL, Shah MR, Hernandez AF, Braunwald E, Redfield MM; NHLBI Heart Failure Clinical Research Network. Low-dose dopamine or low-dose nesiritide in acute heart failure with renal dysfunction: the ROSE acute heart failure randomized trial. JAMA. 2013 Dec 18;310(23):2533-43. doi: 10.1001/jama.2013.282190. PMID 24247300
- [Background] Shchekochikhin D, Lindenfeld J, Schrier R. Increased Spironolactone in Advanced Heart Failure: Effect of Doses Greater than 25 mg/Day on Plasma Potassium Concentration. Cardiorenal Med. 2013 Apr;3(1):1-6. doi: 10.1159/000346447. Epub 2013 Jan 30. PMID 23801997
- [Background] Eng M, Bansal S. Use of natriuretic-doses of spironolactone for treatment of loop diuretic resistant acute decompensated heart failure. Int J Cardiol. 2014 Jan 1;170(3):e68-9. doi: 10.1016/j.ijcard.2013.11.023. Epub 2013 Nov 12. No abstract available. PMID 24268982